CLINICAL TRIAL: NCT04147481
Title: Effects of Abdominal Nerve Block on Postoperative Recovery in Patients Undergoing Gastrointestinal Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Yi Liu (Other)
Responsible Party: Sponsor-Investigator, Yi Liu, Attending doctor, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PLAGHAOC1901
Record Dates: First submitted 2019-10-19; First posted 2019-11-01 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Colon Cancer; Rectal Cancer; Gastric Cancer
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms; Stomach Neoplasms | interventions — Anesthetics, Local; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group Abdominal Nerve Block (Experimental): surgical under general anesthesia combined with transversus abdominis plane block (TAPB) and/or rectus sheath block (RSB) with 0.2% ropivacaine
  Interventions: Other: Group Abdominal Nerve Block with local anesthetics
- Group control (Placebo Comparator): surgical under general anesthesia combined with transversus abdominis plane block (TAPB) and/or rectus sheath block (RSB) with 0.9% saline.
  Interventions: Other: Group Abdominal Nerve Block with saline

INTERVENTIONS:
Other: Group Abdominal Nerve Block with local anesthetics — surgical under general anesthesia combined with transversus abdominis plane block (TAPB) and/or rectus sheath block (RSB) with 0.2% ropivacaine
  Arms: Group Abdominal Nerve Block
Other: Group Abdominal Nerve Block with saline — surgical under general anesthesia combined with transversus abdominis plane block (TAPB) and/or rectus sheath block (RSB) with not 0.2% ropivacaine but 0.9% saline.
  Arms: Group control

SUMMARY:
To explore the effect of general anesthesia combined with transversus abdominis plane block (TAPB) and/or rectus sheath block (RSB) on the recovery of patients with gastrointestinal tumor after surgical treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 80 years.
2. ASA 1-3.
3. Clinical diagnosis of gastric carcinoma and colorectal cancer without metastasis.
4. Surgery for gastrointestinal surgery.

Exclusion Criteria:

1. Patients and their family members refuse to accept the clinical trial;
2. Complicated with acute cholangitis, gastrointestinal bleeding or ascites, etc.;
3. Hepatic encephalopathy, psychosis or neuropathy;
4. Body weight for acid-base and electrolyte imbalances, endotoxemia, and cachexia decreased by more than 2% or 5% in the past 2 months or 6 months.
5. Uncontrolled hypertentsion, coronary heart disease, diabetes.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-10-21 (Actual); Primary Completion 2020-10-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative chronic pain | 6 month after operation
  The incidence of chronic pain 6 month after operation

SECONDARY OUTCOMES:
Bedridden time | The postoperative duration up to 15 days
  Postoperative bedridden time
Fasting time | The postoperative duration up to 15 days
  Postoperative fasting time
Gastrointestinal decompression | The postoperative duration up to 15 days
  Time of gastrointestinal decompression

OTHER OUTCOMES:
The numeric rating scale of postoperative pain | Within 7 days after surgery
  The numerical rating scale (0-10) of posteoperaitve acute pain. If the NRS was larger than 4, we must take emergency action, including pressuring patient controlled analgesia pump, giving other analgesics.

CONTACTS AND LOCATIONS:
Overall Officials: Yi Liu, MD, Study Chair — the Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Haidian, China